CLINICAL TRIAL: NCT06612008
Title: Superimposition of Intra-oral Scans in Mandibular Advancement Device (MAD) Therapy for Obstructive Sleep Apnea
Brief Title: Superimposition of Intra-oral Scans in MAD Therapy for OSA
Acronym: SIMT-OSA
Status: Not yet recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Principal Investigator, Jan de lange, Prinicipal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: 202401
Record Dates: First submitted 2024-09-09; First posted 2024-09-25 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Obstructive Sleep Apnea Syndrome; Oral Appliance Therapy; Mandibular Advancement Device
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stepwise titration: Patients will receive a MAD with an individualized stepwise titration protocol. Initially, the device is set at 60% advancement of the maximum protrusion. Over the first 3 months, the advancement is adjusted incrementally (to 75% or 90%) based on subjective improvement in OSA symptoms and side effects. If side effects occur, the advancement is decreased.
  Interventions: Device: Mandibular Advancement Device
- Personalized titration: Patients will receive a MAD set to baseline settings. Instead of following a standard titration process, personalized titration will use both objective data and subjective patient feedback to determine the optimal advancement. This approach takes into account individual factors such as the patient's oral anatomy, sleep study results, and specific symptoms. The goal is to achieve a personalized, optimal setting that maximizes symptom improvement and comfort.
  Interventions: Device: Mandibular Advancement Device

INTERVENTIONS:
Device: Mandibular Advancement Device — MADs are custom-fitted oral appliances designed to reposition the mandible (lower jaw) forward during sleep, which helps to keep the airway open by preventing upper airway collapse.

SUMMARY:
Obstructive Sleep Apnea (OSA) affects quality of life and health. Mandibular Advancement Devices (MAD) can help with OSA but may cause dental and jaw changes. This study uses a new 3D scanning method to track these changes and compare two adjustment methods for MAD to find the best approach for patients.

Goals:

1. To track dental and jaw changes in OSA patients using 3D scans.
2. To assess the impact of MAD on quality of life and cognitive function.

Study Details:

The aim of the study is to follow OSA patients at multiple centers over several years, comparing two MAD adjustment methods. Participants will undergo routine fitting and imaging.

Outcome:

The study aims to reduce dental and jaw changes and to improve MAD treatment and patient outcomes.

DETAILED DESCRIPTION:
Rationale: Obstructive Sleep Apnea (OSA) significantly reduces quality of life and increases the risk of severe health issue. While Mandibular Advancement Devices (MAD) are effective in managing OSA symptoms, they often introduce undesirable dental and skeletal changes, which can have a negative impact on patient satisfaction. Recognizing this issue, this study hypothesizes that using an innovative 3D superimposition technique to track these changes will allow to compare two different titration protocols more precisely and determine the optimal approach for various patient groups. By identifying the most effective titration protocol, the aim is to enhance treatment adherence and treatment success, addressing a critical gap in existing literature and significantly improving patient outcomes in OSA treatment.

Objective:

1. Investigate dental and skeletal changes in OSA patients undergoing MAD treatment using an innovative 3D superimposition technique.
2. Assess the impact of MAD treatment on quality of life (QoL) and cognitive function.

Study design: A prospective multicentre observational cohort study will be conducted, involving four screening points: at the study's onset and during the first, second, and third annual follow-up assessments. This investigation will involve two patient cohorts undergoing different titration approaches: orthodontic titration and another commonly used titration protocol.

Study population: The study will include adults with mild to moderate OSA who will undergo MAD treatment.

Intervention: Participants will be fitted with a MAD as part of their routine clinical care. The intervention involves the collection of baseline intra-oral scans (IOS), lateral cephalograms (LCR), orthopantomograms (OPT), and a collection of orthodontic parameters. These assessments will be repeated at each follow-up appointment.

Main study parameters/endpoints:

1. Dental and skeletal changes tracked over time using intra-oral scans (IOS), lateral cephalograms (LCR), orthopantomograms (OPT), and complete orthodontic evaluations.
2. Changes in quality of life (QoL) and cognitive function assessed through validated questionnaires.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will experience the routine procedure of MAD fitting and imaging assessments. The study's positive outcomes encompass advancing the knowledge of the enduring impacts of MAD treatment on oral health. Participants will not incur any additional risks by engaging in this research, as it solely involves additional routine diagnostic procedures. The study is group-related, focusing on OSA patients undergoing MAD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Patients with a diagnosis of OSA
* Patients with an apnea-hypopnea index (AHI) of 5 until 30 events per hour
* Patients initially treated with MAD

Exclusion Criteria:

* Patients under 18 years of age
* Patients without a diagnosis of mild to moderate OSA
* Patients undergoing other treatments for OSA
* Patients previously undergone MAD treatment (this also includes over the counter boil and bite MADs)
* Patients diagnosed with central sleep apnea
* Patients undergoing orthodontic treatment (e.g. braces)
* Pregnant patients
* Patients with craniofacial anomalies or syndromes (e.g., Treacher-Collins, Down, Pierre-Robin, Marfan),
* Patients undergoing cancer treatment with chemotherapy or radiation
* Patients with a history of maxillofacial surgery
* Patients with select dental conditions like severe periodontal disease, temporomandibular joint disease, insufficient dentition to support appliance retention in the mouth
* Patients who use bone resorption inhibitors (such as bisphosphonates, calcitonin, SERMs) or the prolonged use, ≥ 6 months of corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants of the research will be recruited from the Department of Oral and Maxillofacial Surgery at 'Isala Hospital Zwolle' and from the orthodontic practice 'Orthodontisten Heemstede', both located in the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Dental occlusal measurements | Baseline; Year 1; Year 2; Year 3
  * Overbite (mm): the vertical overlap of the upper and lower teeth.
  * Overjet (mm): the horizontal overlap of the upper and lower teeth.
  * Maximal protrusion (mm): the most protrusive position of the mandible, independent of tooth contact.
  * Maximal retrusion (mm): the most retrusive position of the mandible, independent of tooth contact.
  * Protrusive range (mm): the distance between the most protrusive and most retrusive position of the mandible.
  * Maximal mouth opening (mm): the maximum distance between the upper and lower incisors when the mouth is fully opened.
Molar and canine relationships | Baseline; Year 1; Year 2; Year 3
  * Molar relationships (in premolar width equivalents): the relative position of the upper and lower molars.
  * Canine relationships (in premolar width equivalents): the relative position of the upper and lower canines.
History of orthodontic treatment | Baseline; Year 1; Year 2; Year 3
  • Previous orthodontic treatment (braces/ premolar extractions)

SECONDARY OUTCOMES:
Cephalometric dentofacial measurements | Baseline; Year 1; Year 2; Year 3
  • Dentofacial profile: Pro- and inclination (degrees)
  • Sagittal facial projection: SNA (degrees), SNB (degrees), and ANB (degrees)
Cephalometric facial and mandibular measurements | Baseline; Year 1; Year 2; Year 3
  • Facial height and divergence: Ar-Go⌃Me (mm), S-N⌃Ar (mm), Na-Me (mm), MP⌃S-Na (mm), and S-Go (mm)
  • Mandibular dimensions: Go-Gn (mm) and Ar-Go (mm)
  • Mandibular plane and hyoid point: MP-Hy (mm)
  • Hyoid point and posterior pharyngeal wall: Hy-PAS (mm)
Cephalometric ratios and divergence | Baseline; Year 1; Year 2; Year 3
  • Facial height and divergence: Ar-Go/N-Me (%)

OTHER OUTCOMES:
Quality of Life (QoL) | Baseline; Year 1; Year 2; Year 3
  * Assessment Tool: Epworth Sleepiness Scale (ESS)
  * Measurement Parameters: Daytime sleepiness, fatigue levels, and overall life satisfaction related to sleep quality
Cognitive Function | Baseline; Year 1; Year 2; Year 3
  * Assessment Tool: Mini-Mental State Examination (MMSE)
  * Measurement Parameters: Attention, memory, orientation and executive function
Sleep Quality | Baseline; Year 1; Year 2; Year 3
  * Assessment Tool: Pittsburgh Sleep Quality Index (PSQI)
  * Measurement Parameters: Sleep latency, duration, efficiency, disturbances, and overall sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: J. de Lange, Prof. Dr., Principal Investigator — Amsterdam University Medical Center; J.P.T.F. Ho, Dr., Principal Investigator — Amsterdam University Medical Center; N.C.W. van der Kaaij, Dr., Principal Investigator — Amsterdam University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Ruiter MHT, Aarab G, de Vries N, Lobbezoo F, de Lange J. A stepwise titration protocol for oral appliance therapy in positional obstructive sleep apnea patients: proof of concept. Sleep Breath. 2020 Sep;24(3):1229-1236. doi: 10.1007/s11325-020-02045-w. Epub 2020 Mar 11. PMID 32162278
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7426292/